CLINICAL TRIAL: NCT03218787
Title: A Safety Evaluation of 3-month Dual Antiplatelet Therapy in Subjects at High Risk of Bleeding Undergoing Percutaneous Coronary Intervention With XIENCE.
Brief Title: XIENCE 90: A Safety Evaluation of 3-month DAPT After XIENCE Implantation for HBR Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-308
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Lesions
Keywords: Coronary Artery Lesions; XIENCE; Dual Antiplatelet Therapy (DAPT); Reduced DAPT; Risk of bleeding; Drug-eluting stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- XIENCE (Experimental): Subjects will receive XIENCE family stents and if a subject was DAPT compliant and event free, then took 3 month DAPT, following with aspirin mono-therapy until 12 month
  Interventions: Device: XIENCE; Drug: DAPT

INTERVENTIONS:
Device: XIENCE — Subjects who received XIENCE family stent systems will be included.
Drug: DAPT — 3-month clear subjects who receive 3-month DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days.
  Subject who are "3-month clear" will discontinue P2Y12 inhibitor after 3-month visit, but continue taking aspirin through 12-month follow-up. Subjects who are not eligible for early P2Y12 inhibitor discontinuation will be treated per site standard of care.
  Other Names: Dual antiplatelet therapy

SUMMARY:
XIENCE 90 study is a prospective, single arm, multi-center, open label trial to evaluate the safety of 3-month dual antiplatelet therapy (DAPT) in subjects at high risk of bleeding (HBR) undergoing percutaneous coronary intervention (PCI) with the approved XIENCE family of coronary drug-eluting stents.

The XIENCE family stent systems include commercially approved XIENCE Xpedition Everolimus Eluting Coronary Stent System (EECSS), XIENCE Alpine EECSS, XIENCE PRO^X EECSS [rebrand of the XIENCE Xpedition Stent System and is only available outside of the United States (OUS)], XIENCE PRO^A EECSS (rebrand of the XIENCE Alpine Stent System and is only available OUS) and XIENCE Sierra EECSS of coronary drug-eluting stents.

DETAILED DESCRIPTION:
A. Primary Objective:

To show non-inferiority of the primary endpoint of all death or all MI (modified ARC) from 3 to 12 months following XIENCE implantation in HBR subjects treated with 3-month DAPT compared to a historical control after propensity score adjustment.

B. Secondary Objective:

* To show superiority of the major secondary endpoint of major bleeding (Bleeding Academic Research Consortium [BARC] type 2-5) from 3 to 12 months following XIENCE implantation in HBR subjects treated with 3-month DAPT compared to a historical control after propensity score adjustment.
* To evaluate stent thrombosis (ARC definite/probable) from 3 to 12 months following XIENCE implantation in HBR subjects treated with 3-month DAPT against a performance goal (PG).

All registered subjects will be followed at 3, 6 and 12 months post index procedure.

The data collected from this study will be compared with the historical control of non-complex HBR subjects treated with standard DAPT duration of up to 12 months from the XIENCE V USA study, which is a US post-approval study to evaluate the safety of XIENCE V EECSS in "all-comer" population under real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is considered at high risk for bleeding (HBR), defined as meeting one or more of the following criteria at the time of registration and in the opinion of the referring physician, the risk of major bleeding with > 3-month DAPT outweighs the benefit:

   1. ≥ 75 years of age.
   2. Clinical indication for chronic (at least 6 months) or lifelong anticoagulation therapy.
   3. History of major bleeding which required medical attention within 12 months of the index procedure.
   4. History of stroke (ischemic or hemorrhagic).
   5. Renal insufficiency (creatinine ≥ 2.0 mg/dl) or failure (dialysis dependent).
   6. Systemic conditions associated with an increased bleeding risk (e.g. hematological disorders, including a history of or current thrombocytopenia defined as a platelet count <100,000/mm^3, or any known coagulation disorder associated with increased bleeding risk).
   7. Anemia with hemoglobin < 11g/dl.
2. Subject must be at least 18 years of age.
3. Subject or a legally authorized representative must provide written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site prior to any study related procedure.
4. Subject is willing to comply with all protocol requirements, including agreement to stop taking P2Y12 inhibitor at 3 months, if eligible per protocol.
5. Subject must agree not to participate in any other clinical trial for a period of one year following the index procedure.

Angiographic Inclusion Criteria

1. Up to three target lesions with a maximum of two target lesions per epicardial vessel. Note:

   * The definition of epicardial vessels means left anterior descending coronary artery (LAD), left circumflex coronary artery (LCX) and right coronary artery (RCA) and their branches. For example, the patient must not have >2 lesions requiring treatment within both the LAD and a diagonal branch in total.
   * If there are two target lesions within the same epicardial vessel, the two target lesions must be at least 15 mm apart per visual estimation; otherwise this is considered as a single target lesion.
2. Target lesion ≤ 32 mm in length by visual estimation.
3. Target lesion must be located in a native coronary artery with visually estimated reference vessel diameter between 2.25 mm and 4.25 mm.
4. Exclusive use of XIENCE family of stent systems during the index procedure.
5. Target lesion has been treated successfully, which is defined as achievement of a final in-stent residual diameter stenosis of <20% with final TIMI-3 flow assessed by online quantitative angiography or visual estimation, with no residual dissection NHLBI grade ≥ type B, and no transient or sustained angiographic complications (e.g., distal embolization, side branch closure), no chest pain lasting > 5 minutes, and no ST segment elevation > 0.5 mm or depression lasting > 5 minutes.

General Exclusion Criteria

1. Subject with an indication for the index procedure of acute ST-segment elevation MI (STEMI).
2. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, P2Y12 inhibitors (clopidogrel/prasugrel/ticagrelor), everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
3. Subject with implantation of another drug-eluting stent (other than XIENCE) within 9 months prior to index procedure.
4. Subject has a known left ventricular ejection fraction (LVEF) <30%.
5. Subject judged by physician as inappropriate for discontinuation from P2Y12 inhibitor use at 3 months, due to another condition requiring chronic P2Y12 inhibitor use.
6. Subject with planned surgery or procedure necessitating discontinuation of P2Y12 inhibitor within 3 months following index procedure.
7. Subject with a current medical condition with a life expectancy of less than 12 months.
8. Subject intends to participate in an investigational drug or device trial within 12 months following the index procedure.
9. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

   Note: Female patients of childbearing potential should be instructed to use safe contraception (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches, hormonal vaginal devices, injections with prolonged release.) It is accepted, in certain cases, to include subjects having a sterilised regular partner or subjects using a double barrier contraceptive method. However, this should be explicitly justified in special circumstances arising from the study design, product characteristics and/or study population
10. Subject is part of a vulnerable population, defined as subject whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples of populations which may contain vulnerable subjects include: individuals with lack of or loss of autonomy due to immaturity or through mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, and those incapable of giving informed consent. Other vulnerable subjects include, for example, members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces, and persons kept in detention.
11. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.

Angiographic Exclusion Criteria

1. Target lesion is in a left main location.
2. Target lesion is located within an arterial or saphenous vein graft.
3. Target lesion is restenotic from a previous stent implantation.
4. Target lesion is a total occluded lesion (TIMI flow 0).
5. Target lesion contains thrombus as indicated in the angiographic images (per SYNTAX score thrombus definition).
6. Target lesion is implanted with overlapping stents, whether planned or for bailout.

Note: If there is more than one target lesion, all target lesions must satisfy the angiographic eligibility criteria. Non-target lesion (i.e., lesions that do not meet the angiographic criteria listed above) treatments are not allowed during the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2047 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, Principal Investigator — Abbott Medical Devices
Locations (101):
- United States (101):
  - Huntsville Hospital (Heart Center Research LLC), Huntsville, Alabama
  - Scottsdale Healthcare Hospitals (d/b/a HonorHealth - HonorHealth Research Institute), Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - John Muir Health Concord, Concord, California
  - Washington Hospital (Mission Cardiovascular Research Institute), Fremont, California
  - Scripps Memorial Hospital/Prebys Cardiovascular Institute, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Sharp Grossmont Hospital (La Mesa Cardiac Center), San Diego, California
  - Sharp Memorial Hospital / San Diego Cardiac Center, San Diego, California
  - Santa Barbara Cottage Hospital/Sansum Clinic, Santa Barbara, California
  - Torrance Memorial Medical Center, Torrance, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Medstar Washington Hospital, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - Clearwater Cardiovasular Consultants, Clearwater, Florida
  - Morton Plant Mease Healthcare System, Clearwater, Florida
  - North Florida Regional / The Cardiac and Vascular Institute, Gainesville, Florida
  - St. Vincent's Medical Center (St. Vincent's Healthcare), Jacksonville, Florida
  - Tallahassee Memorial Hospital / Tallahassee Research Institute, Inc., Tallahassee, Florida
  - University Health, INC/University Cardiology Associates, LLC, Augusta, Georgia
  - Augusta Medical Center, Augusta, Georgia
  - Atlanta Veterans Affairs Medical Center, Decatur, Georgia
  - North Georgia Heart Foundation, Inc., Gainesville, Georgia
  - St. John's Hospital, Springfield, Illinois
  - Elkhart General Hospital/Midwest Cardiology Research & Education Foundation, Elkhart, Indiana
  - Franciscan Physician Network-Indiana Heart Physicians, Indianapolis, Indiana
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas/Via Christi Regional Medical, Wichita, Kansas
  - Kansas Heart Hospital (Cardiovascular Research Institute of Kansas), Wichita, Kansas
  - University of Kentucky/Gill Heart and Vascular Institute, Lexington, Kentucky
  - Baptist Health Louisville/Louisville Cardiology, Louisville, Kentucky
  - Eastern Maine Medical Center/One Northeast Drive, Bangor, Maine
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic/Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - McLaren Bay Region, Bay City, Michigan
  - St John Hospital & Medical Center, Detroit, Michigan
  - Genesys Regional Medical Center (Regional Cardiology Associates), Grand Blanc, Michigan
  - Western Michigan University Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - MidMichigan Medical Center Midland, Midland, Michigan
  - Traverse Heart and Vascular Munson Medical Center, Traverse City, Michigan
  - St. Joseph Mercy Hospital (Michigan Heart), Ypsilanti, Michigan
  - Abbott Northwestern Hospital (Minneapolis Heart Institute Foundation), Minneapolis, Minnesota
  - CentraCare, Saint Cloud, Minnesota
  - St Dominic-Jackson Memorial Hospital (Jackson Heart Clinic), Jackson, Mississippi
  - North Mississippi Medical Center (Cardiology Associates Research), Tupelo, Mississippi
  - Boone Hospital Center (Missouri Cardiovascular Specialists), Columbia, Missouri
  - St. Luke's Hospital/Mid America Heart Institute, Kansas City, Missouri
  - Washington University School of Medicine Barnes Jewish Hospital, St Louis, Missouri
  - St. Patrick Hospital International Heart Institute of Montana Foundation, Missoula, Montana
  - Bryan Local General Hospital (Bryan Medical Center East), Lincoln, Nebraska
  - Our Lady of Lourdes/Cardiovascular Associates of the Delaware Valley (The Heart House), Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - St. Joseph's Hospital Health Center, East Syracuse, New York
  - New York - Presbyterian Queens Lang Research Center, Flushing, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital - Weill Cornell, New York, New York
  - Lenox Hill Hospital (Northwell)/ Feinstein Institute, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - The Presbyterian Hospital (d/b/a Novant Health Heart and Vascular Institute) Novant Health Clinical Research, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center (Wake Forest University Health Sciences)/Medical Center Boulevard, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cardiovascular Research Center, LLC (Mercy Health St. Vincent Medical Center LLC), Toledo, Ohio
  - Integris Baptist Medical Center/Integris Cardiovascular Physicians, LLC, Oklahoma City, Oklahoma
  - Hillcrest Medical Center (Oklahoma Heart Institute), Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Hamot/Medicor Associates, Inc.,, Erie, Pennsylvania
  - Harrisburg Hospital/Pinnacle Health Cardiovascular Institute, Inc., Harrisburg, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Penn Presbyterian Medical Center/Penn Heart and Vascular Pavilion,, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Wyomissing, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Clinical Research, Anderson, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Turkey Creek Medical Center (Knoxville HMA Cardiology, LLC), Knoxville, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Centennial Medical Center (TriStar Centennial Medical Center), Nashville, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Memorial Hermann-Hermann Hospital/UTHealth, Houston, Texas
  - Texas Tech University Health (University Medical Center), Lubbock, Texas
  - East Texas Medical Center, Tyler, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Inova Fairfax Hospital/Inova Heart and Vascular Institute, Falls Church, Virginia
  - Mary Washington Hospital/Virginia Cardiovascular Consultants, Fredericksburg, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Charleston Area Medical Center Memorial Division, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valgimigli M, Cao D, Angiolillo DJ, Bangalore S, Bhatt DL, Ge J, Hermiller J, Makkar RR, Neumann FJ, Saito S, Picon H, Toelg R, Maksoud A, Chehab BM, Choi JW, Campo G, De la Torre Hernandez JM, Kunadian V, Sardella G, Thiele H, Varenne O, Vranckx P, Windecker S, Zhou Y, Krucoff MW, Ruster K, Zheng Y, Mehran R; XIENCE 90 and XIENCE 28 Investigators. Duration of Dual Antiplatelet Therapy for Patients at High Bleeding Risk Undergoing PCI. J Am Coll Cardiol. 2021 Nov 23;78(21):2060-2072. doi: 10.1016/j.jacc.2021.08.074. PMID 34794687
- [Derived] Valgimigli M, Cao D, Makkar RR, Bangalore S, Bhatt DL, Angiolillo DJ, Saito S, Ge J, Neumann FJ, Hermiller J, Picon H, Toelg R, Maksoud A, Chehab BM, Wang LJ, Wang J, Mehran R. Design and rationale of the XIENCE short DAPT clinical program: An assessment of the safety of 3-month and 1-month DAPT in patients at high bleeding risk undergoing PCI with an everolimus-eluting stent. Am Heart J. 2021 Jan;231:147-156. doi: 10.1016/j.ahj.2020.09.019. Epub 2020 Oct 6. PMID 33031789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2047 subjects were registered in XIENCE 90 from 101 sites in the US between 19 July, 2017 and 09 August, 2019. The last patient visit was on 04 September, 2020.
Groups:
- XIENCE: XIENCE: Subjects will receive XIENCE family stents and if a subject was DAPT compliant and event free, then took 3 month DAPT, following with aspirin mono-therapy until 12 month
  DAPT: 3-month clear subjects who receive 3-month DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days.
  Subject who are "3-month clear" will discontinue P2Y12 inhibitor after 3-month visit, but continue taking aspirin through 12-month follow-up. Subjects who are not eligible for early P2Y12 inhibitor discontinuation will be treated per site standard of care.
Period: Overall Study
Arm/Group | XIENCE
Started | 2047
Completed | 1841
Not Completed | 206
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 72
Not completed — Physician Decision | 11
Not completed — Death | 111

BASELINE CHARACTERISTICS:
Arm/Group | XIENCE
Number analyzed (Participants) | 2047
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.10 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 726
  Male | 1321
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 45
  Black or African American | 125
  Hispanic or Latino | 57
  Native Hawaiian or Pacific Islander | 6
  White | 1804
  Did not wish to disclose | 55
  Not available | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2047
Chronic anticoagulant [Count of Participants; unit: Participants] | 836

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Rate of All Death or All Myocardial Infarction (MI)(Modified Academic Research Consortium [ARC]), by Propensity Score Quintiles
Description: All death: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease should be classified as cardiac.
  MI (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block, development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI
  * Spontaneous MI: CK-MB > URL or Troponin > URL with baseline value < UR
  The propensity score for each individual was calculated using a logistic regression model that included the study group as the outcome & the baseline demographic, clinical and procedural covariates as the predictors
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Percentage of participants
  Adjusted Overall Rate | 5.4
  Q1: number analyzed (Participants) | 104
  Q1 | 6.7
  Q2: number analyzed (Participants) | 225
  Q2 | 4.0
  Q3: number analyzed (Participants) | 361
  Q3 | 3.6
  Q4: number analyzed (Participants) | 446
  Q4 | 5.8
  Q5: number analyzed (Participants) | 536
  Q5 | 6.9

2. Secondary Outcome: Percentage of Participants With Major Bleeding Rate by Bleeding Academic Research Consortium (BARC) Type 2-5, by Propensity Score Quintiles
Description: * Type 2: Any overt, actionable sign of hemorrhage
  * Type 3a: Overt bleeding plus Hb drop of 3 to < 5g/dL;Any transfusion with overt bleeding
  * Type 3b: Overt bleeding plus Hb drop ≥ 5 g/dL;Cardiac tamponade;Bleeding requiring surgical intervention for control;Bleeding requiring IV vasoactive agents
  * Type 3c: ICH; Subcategories confirmed by autopsy/imaging/lumbar puncture;Intraocular bleed compromising vision
  * Type 4: CABG-related bleeding: Perioperative intracranial bleeding within 48h;Reoperation after closure of sternotomy for the purpose of controlling bleeding;Transfusion of ≥ 5 U whole blood or packed RBC within 48h;Chest tube output ≥ 2L within 24h
  * Type 5: Fatal bleeding
  The propensity score for each individual was calculated using a logistic regression model that included the study group as the outcome & the baseline demographic, clinical and procedural covariates as the predictors.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1629
Percentage of participants
  Adjusted Overall Rate | 5.1
  Q1: number analyzed (Participants) | 102
  Q1 | 3.9
  Q2: number analyzed (Participants) | 221
  Q2 | 2.7
  Q3: number analyzed (Participants) | 353
  Q3 | 5.4
  Q4: number analyzed (Participants) | 435
  Q4 | 6.0
  Q5: number analyzed (Participants) | 518
  Q5 | 7.7

3. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable)
Description: Definite stent thrombosis:
  Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation.
  Probable stent thrombosis:
  Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases:
  * Any unexplained death within the first 30 days
  * Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1635
Participants | 4

4. Secondary Outcome: Number of Participants With All Death, Cardiac Death, Vascular Death, Non-cardiovascular Death
Description: All Death:
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  Cardiac death:
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death:
  Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death:
  Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 54

5. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI) and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: All Myocardial Infarction (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI:
    * Within 48h after PCI: CK-MB >3 x URL or Troponin > 3 x URL with baseline value < URL
    * Within 72h after CABG: CK-MB >5 x URL or Troponin > 5 x URL with baseline value < URL
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
  TV-MI: All infarcts that cannot be clearly attributed to a vessel other than the target vessel will be considered related to the target vessel.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 48

6. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: Cardiac death:
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  MI (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI:
    * Within 48h after PCI: CK-MB >3 x URL or Troponin > 3 x URL with baseline value < URL
    * Within 72h after CABG: CK-MB >5 x URL or Troponin > 5 x URL with baseline value < URL
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 67

7. Secondary Outcome: Number of Participants With All Stroke, Ischemic Stroke and Hemorrhagic Stroke
Description: An acute symptomatic episode of neurological dysfunction attributed to a vascular cause lasting more than 24 hours or lasting 24 hours or less with a brain imaging study or autopsy showing new infarction.
  * Ischemic Stroke: An acute symptomatic episode of focal cerebral, spinal, or retinal dysfunction caused by an infarction of central nervous system tissue.
  * Hemorrhagic Stroke: An acute symptomatic episode of focal or global cerebral or spinal dysfunction caused by a non-traumatic intraparenchymal, intraventricular, or subarachnoid hemorrhage.
  * Undetermined Stroke: A stroke with insufficient information to allow categorization as ischemic or hemorrhagic.
  * Pharmacologic, i.e., thrombolytic drug administration, or Non-pharmacologic, i.e., neurointerventional procedure (e.g., intracranial angioplasty)
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1624
Participants | 21

8. Secondary Outcome: Number of Participants With Clinically-indicated Target Lesion Revascularization (CI-TLR)
Description: Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not clinically indicated by the investigator prior to repeat angiography.
  Clinically Indicated [CI] Revascularization:
  A revascularization is considered clinically indicated if angiography at follow-up shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  * A positive history of recurrent angina pectoris, presumably related to the target vessel;
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  * Abnormal results of any invasive functional diagnostic test
  * A TLR/TVR with a diameter stenosis ≥70% in the absence of the above mentioned ischemic signs or symptoms.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 16

9. Secondary Outcome: Number of Participants With Clinically-indicated Target Vessel Revascularization (CI-TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
  A revascularization is considered clinically indicated if angiography at follow-up shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  * A positive history of recurrent angina pectoris, presumably related to the target vessel;
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  * Abnormal results of any invasive functional diagnostic test (e.g., Doppler flow velocity reserve, fractional flow reserve);
  * A TVR with a diameter stenosis ≥70% in the absence of the above mentioned ischemic signs or symptoms.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 26

10. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: TLF is defined as a composite of all cardiac death, myocardial infarction attributed to target vessel or clinically-indicated TLR.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 66

11. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, Composite of Cardiac Death, TV-MI and CI-TVR)
Description: TVF is defined as a composite of cardiac death, MI attributed to target vessel, clinically-indicated TLR, or clinically-indicated TVR, non-TLR.
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1672
Participants | 70

12. Secondary Outcome: Number of Participants With Major Bleeding Defined by the Bleeding Academic Research Consortium (BARC) Type 3-5
Description: Bleeding per Bleeding Academic Research Consortium (BARC) adjudicated definitions are as follows:
  * Type 3a: Overt bleeding plus Hemoglobin(Hb) drop of 3 to < 5 g/dL; Any transfusion with overt bleeding
  * Type 3b: Overt bleeding plus Hb drop ≥ 5 g/dL; Cardiac tamponade; Bleeding requiring surgical intervention for control; Bleeding requiring IV vasoactive agents
  * Type 3c: Intracranial hemorrhage;Subcategories confirmed by autopsy or imaging or lumbar puncture; Intraocular bleed compromising vision
  * Type 4: CABG-related bleeding: Perioperative intracranial bleeding within 48 h; Reoperation after closure of sternotomy for the purpose of controlling bleeding; Transfusion of ≥ 5 U whole blood or packed red blood cells within a 48-h period; Chest tube output ≥ 2L within a 24-h period
  * Type 5: Fatal bleeding
  * Type 5a: Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious
  * Type 5b: Definite fatal bleeding;overt bleeding or autopsy or imaging confirmation
Time Frame: From 3 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1629
Participants | 41

ADVERSE EVENTS:
Time Frame: 1 Year
Groups:
- XIENCE: Subjects will receive XIENCE family stent systems and 3-month DAPT
  XIENCE: Subjects will receive XIENCE family stents and if a subject was DAPT compliant and event free, then took 3 month DAPT, following with aspirin mono-therapy until 12 month
  DAPT: 3-month clear subjects who receive 3-month DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days.
  Subject who are "3-month clear" will discontinue P2Y12 inhibitor after 3-month visit, but continue taking aspirin through 12-month follow-up. Subjects who are not eligible for early P2Y12 inhibitor discontinuation will be treated per site standard of care.
Arm/Group | XIENCE
All-Cause Mortality (participants affected / at risk) | 115/2047
Serious Adverse Events (participants affected / at risk) | 898/2047
Other Adverse Events (participants affected / at risk) | 129/2047
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE (N=2047)
Anaemia (Blood and lymphatic system disorders) | 60 (62)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 14 (15)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 4 (4)
Angina pectoris (Cardiac disorders) | 146 (180)
Angina unstable (Cardiac disorders) | 5 (5)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 4 (4)
Arrhythmia (Cardiac disorders) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 101 (116)
Atrial flutter (Cardiac disorders) | 15 (16)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 5 (5)
Atrioventricular block second degree (Cardiac disorders) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 20 (21)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 16 (16)
Cardiac disorder (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 14 (15)
Cardiac failure acute (Cardiac disorders) | 11 (12)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 87 (109)
Cardiac perforation (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 8 (9)
Cardiomyopathy (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 15 (15)
Coronary artery dissection (Cardiac disorders) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 6 (6)
Mitral valve stenosis (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 56 (65)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 6 (6)
Pericarditis (Cardiac disorders) | 2 (2)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 6 (6)
Sinus arrest (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 6 (6)
Tachycardia (Cardiac disorders) | 3 (3)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (3)
Ventricular tachycardia (Cardiac disorders) | 12 (12)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 3 (4)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Retinoschisis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Colonic polyp (Gastrointestinal disorders) | 4 (4)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 43 (46)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 7 (7)
Haematochezia (Gastrointestinal disorders) | 9 (9)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 3 (3)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Melaena (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (3)
Oesophageal hypomotility (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 7 (7)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 3 (3)
Small intestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 8 (8)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (7)
Volvulus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Accidental death (General disorders) | 1 (1)
Asthenia (General disorders) | 9 (10)
Catheter site haematoma (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 2 (2)
Chest discomfort (General disorders) | 4 (4)
Chest pain (General disorders) | 6 (6)
Death (General disorders) | 9 (9)
Device capturing issue (General disorders) | 1 (1)
Device malfunction (General disorders) | 2 (2)
Feeling hot (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Injection site extravasation (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 37 (40)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (3)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 3 (6)
Ulcer (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
Antiphospholipid syndrome (Immune system disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Pancreas transplant rejection (Immune system disorders) | 1 (2)
Sarcoidosis (Immune system disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arteritis infective (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 6 (6)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 22 (22)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Clostridium difficile sepsis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Eye infection staphylococcal (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 4 (4)
Gastroenteritis (Infections and infestations) | 6 (6)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Lobar pneumonia (Infections and infestations) | 5 (6)
Localised infection (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 14 (14)
Parotitis (Infections and infestations) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 47 (52)
Pneumonia primary atypical (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 11 (12)
Septic embolus (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 7 (7)
Staphylococcal abscess (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 2 (3)
Tooth abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 22 (24)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4)
Wound abscess (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Complications of transplanted pancreas (Injury, poisoning and procedural complications) | 1 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Dialysis related complication (Injury, poisoning and procedural complications) | 2 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 20 (20)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (3)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3)
Foreign body (Injury, poisoning and procedural complications) | 2 (2)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 8 (8)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 2 (2)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (3)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 (4)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 6 (6)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 10 (10)
Wound haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 3 (3)
Cardiac monitoring (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Occult blood positive (Investigations) | 1 (1)
Troponin increased (Investigations) | 4 (4)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 10 (10)
Hypoglycaemia (Metabolism and nutrition disorders) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Malignant splenic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 9 (9)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 40 (42)
Cervical cord compression (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4)
Dementia (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Diplegia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Dysarthria (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 6 (6)
Essential tremor (Nervous system disorders) | 1 (1)
Frontotemporal dementia (Nervous system disorders) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Hypokinesia (Nervous system disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 5 (5)
Mononeuropathy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 5 (5)
Radiculopathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 27 (32)
Toxic encephalopathy (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 12 (12)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (7)
Bladder mass (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 9 (10)
Nephrolithiasis (Renal and urinary disorders) | 4 (4)
Renal artery stenosis (Renal and urinary disorders) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 44 (48)
Renal failure chronic (Renal and urinary disorders) | 10 (10)
Renal haemorrhage (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 4 (4)
Renal mass (Renal and urinary disorders) | 2 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 34 (38)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 (36)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 19 (21)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 18 (18)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5)
Extremity necrosis (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 2 (3)
Haematoma (Vascular disorders) | 13 (13)
Haemorrhage (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 12 (12)
Hypertensive crisis (Vascular disorders) | 8 (8)
Hypertensive emergency (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 26 (27)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 6 (7)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (7)
Peripheral ischaemia (Vascular disorders) | 6 (7)
Peripheral vascular disorder (Vascular disorders) | 2 (3)
Reperfusion injury (Vascular disorders) | 1 (1)
Secondary hypertension (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Steal syndrome (Vascular disorders) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
Venous occlusion (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE (N=2047)
Angina pectoris (Cardiac disorders) | 129 (139)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03218787/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT03218787/SAP_001.pdf